CLINICAL TRIAL: NCT03483649
Title: Randomized, Double Blind, Intravenous, Single Dose, Parallel, 4-arm Comparative Pharmacokinetic, Safety and Immunogenicity Phase I Study of HLX04 Versus US-sourced Avastin®, EU-sourced Avastin®, and CN-sourced Avastin® in Healthy Male Subjects
Brief Title: Pharmacokinetic, Safety and Immunogenicity Phase I Study of HLX04 Versus Avastin® in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX04 HV01
Record Dates: First submitted 2017-11-30; First posted 2018-03-30 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- HLX04 (Experimental)
  Interventions: Drug: HLX04
- United States (US) Avastin® (Active Comparator)
  Interventions: Drug: US-Avastin®
- European Union (EU) Avastin® (Active Comparator)
  Interventions: Drug: EU-Avastin®
- China (CN) Avastin® (Active Comparator)
  Interventions: Drug: CN-Avastin®

INTERVENTIONS:
Drug: HLX04 — HLX04: Supplied as 100 mg/4 mL solution; reconstituted to 100 mL with 0.9% sodium chloride; a single dose of 3 mg/kg will be administered intravenously for 90 minutes.
  Arms: HLX04
Drug: US-Avastin® — US Avastin®: Supplied as 100 mg/4 mL solution; reconstituted to 100 mL with 0.9% sodium chloride; a single dose of 3 mg/kg will be administered intravenously for 90 minutes.
  Arms: United States (US) Avastin®
Drug: EU-Avastin® — EU-Avastin®: Supplied as 100 mg/4 mL solution; reconstituted to 100 mL with 0.9% sodium chloride; a single dose of 3 mg/kg will be administered intravenously for 90 minutes.
  Arms: European Union (EU) Avastin®
Drug: CN-Avastin® — CN-Avastin®: Supplied as 100 mg/4 mL solution; reconstituted to 100 mL with 0.9% sodium chloride; a single dose of 3 mg/kg will be administered intravenously for 90 minutes.
  Arms: China (CN) Avastin®

SUMMARY:
This is a Phase I, randomized, double blind, IV, single dose, 4-arm parallel study to compare the PK, and to evaluate the safety, tolerability and immunogenicity of HLX04, US Avastin®, EU Avastin®, and CN Avastin® in healthy male subjects.

DETAILED DESCRIPTION:
A total of 188 evaluable male subjects are required. Taking into account a dropout rate of approximately 10%, a total of 208 healthy male subjects who meet the required entry criteria will be randomly assigned to one of four treatment groups in a 1:1:1:1 ratio to receive a single IV infusion of HLX04, EU Avastin® or US Avastin®. The first 8 subjects (with at least 2 subjects receiving HLX04) will be dosed as a maximum of 1 subject per day. Prior to administration of study drug to the next subject, the safety findings of the preceding subject must be reviewed by the Principal Investigator. Each subject will be required to remain in the study center for 96 hours after dosing (overnight) for safety evaluation. After the first 8 subjects are evaluated and the experimental drug deemed safe, the Principal Investigator will decide the continuous enrollment in the four parallels according to the Phase I clinical trial unit capability.

The duration of participation for each subject is expected to be approximately120 days starting with a 21 day screening period, followed by administration of study drug and a 99 day follow up period.

After the follow up visit on Day 99, subjects who are confirmed positive for anti drug antibody (ADA) will be followed for 12 months after study drug administration or until 2 consecutive samples are tested negative for ADA.

The start of study is considered the date of the first subject providing informed consent and the end of study will be the last subject's last scheduled visit (Day 99 or early termination). Additional follow up visits for subjects who are positive for ADAs or have ongoing/resolving adverse events (AEs) will be conducted and recorded separately.

Subjects who meet all eligibility criteria and have signed the informed consent form (ICF) will be admitted to the Phase I clinical trial unit the day prior to dosing (Day 1) and will be discharged 96 hours postdose on Day 5. Then after, subjects will be followed up and continue participation in the study on an outpatient basis for further safety assessments, for blood sampling for PK and to test for ADA and neutralizing ADA (NADA) at selected visits.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing to comply with the contraception restrictions for this study (see Section 4.3.3).
2. Subjects who are able and willing to give written informed consent.
3. Subjects who are willing to comply with the study restrictions from screening until end of study.
4. Adult males aged 18 to 50 years inclusive and between 19 and 26 kg/m2 body mass index and body weight ≥ 50 kg and ≤ 80 kg.
5. Subjects who are non smokers or have not used tobacco or nicotine containing products for at least 3 months preceding screening and have less than 5 cigarettes per day smoking history. Subjects must agree to refrain from smoking during days of confinement at the study center.
6. Subjects negative for Hepatitis B surface antigen, Hepatitis C virus antibody, Treponema pallidum antibody, and human immunodeficiency virus antibody tests.
7. Subjects negative for urine drug screen and alcohol tests.
8. Subjects determined healthy by medical history, physical examination, laboratory tests, 12 lead electrocardiogram (ECG), and chest X ray, without any clinically significant abnormality judged by the Investigator.

Exclusion Criteria:

1. History of gastrointestinal, endocrine, pulmonary, hepatic, renal, psychiatric, neurological, cardiovascular, hematological, and metabolic (including known diabetes mellitus) disease or disorder considered as significant by the Investigator.
2. History of any cancer, lymphoma, or leukemia, except basal cell carcinoma of skin after localized cancer is removed.
3. History or current clinically significant atopic allergy, hypersensitivity or allergic reactions including known or suspected clinically relevant drug hypersensitivity to any component of the study drug formulations or comparable drugs.
4. Any disorder that, in the Investigator's opinion, may interfere with the safety of the subject and the study procedures and evaluations.
5. Blood loss or blood donation (including blood components donation) ≥ 400 mL or blood transfusion within 3 months before screening; blood loss or blood donation (including blood components donation) ≥ 200 mL within 1 months before screening.
6. Surgery within the past 8 weeks or surgery planned during the study duration.
7. Poor oral hygiene that may require surgical intervention during the study or any planned dental interventions during the study duration.
8. Live virus vaccination within 4 weeks prior to screening or intention to receive live virus vaccination during the study until the final follow up visit.
9. History of prior exposure to bevacizumab or any anti VEGF or anti VEGF receptor (VEGFR) monoclonal antibodies or proteins (e.g., aflibercept, ramucirumab, lapatinib, and sunitinib).
10. Prior exposure to any other investigational monoclonal antibody within 12 months of study drug administration.
11. Use of any investigational drug in any clinical study within the 3 months prior to first dose administration in this study; or remains on follow up of any clinical study.
12. Any intake of a non steroidal anti inflammatory drug (NSAID) including any dose of aspirin in the last 14 days. NSAIDs are not allowed for the duration of the study. Paracetamol is allowed for pain control if required.
13. Intake of prescribed or over the counter drugs within 28 days of study drug administration or herbal drugs or dietary supplements within 28 days prior to study drug administration.
14. Any persons who are:

    * An employee of the Principal Investigators, study centers, contract research organization (CRO) or the Sponsor.
    * A relative of an employee of the study centers, the Investigators, CRO or the Sponsor.
15. Abnormal ECG with clinical significance judged by the Investigator.
16. Abnormal serum Immunoglobulin G with clinical significance judged by the Investigator.
17. Confirmed positive ADA at screening.
18. Occurrence of acute disease during screening or predose, e.g., acute hepatitis, acute diarrhea.
19. Intake of any product containing alcohol within 24 hours of study drug administration.
20. Subjects with relevant family history of hypertension or abnormal blood pressure at screening or admission to the study center (Day 1):

    * Systolic blood pressure > 140 mmHg
    * Diastolic blood pressure > 90 mmHg.
21. Any inherited predisposition to bleeding or to thrombosis or history of non traumatic hemorrhage (i.e., requiring medical intervention), thromboembolic event or any condition which may increase bleeding risk including clotting disorders, thrombocytopenia (platelet count < 100000/µL) or an international normalized ratio (INR) higher than 1.5.
22. Any clinically significant infection ongoing at screening or admission to the Phase I clinical trial unit.
23. Total cholesterol > 1.5×upper limit of normal or fasting glucose abnormality with clinical significance at screening or admission.
24. History of alcohol abuse or a positive alcohol breath test, history of drug abuse or positive urine drug screen.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2017-10-29 (Actual); Study Completion 2017-10-29 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) | from 0 to day 99
  Area under the concentration time curve of the analyte in serum over the time interval from 0 to the last quantifiable concentration at time "t" [AUC(0-t)]
AUC(0-∞) | from 0 to day 99
  Area under the concentration time curve of the analyte in serum over the time interval from 0 extrapolated to infinity [AUC(0-∞)]

SECONDARY OUTCOMES:
Cmax | from 0 to day 99
  Maximum measured concentration of the analyte in serum (Cmax)
TEAE and SAE | from 0 to day 99
  Treatment emergent adverse events and serious adverse events
tmax | from 0 to day 99
  • Time from dosing to maximum measured concentration (tmax)
t1/2 | from 0 to day 99
  • Terminal half life of the analyte in serum (t1/2)
λz | from 0 to day 99
  • Terminal elimination rate constant (λz)
CL | from 0 to day 99
  • Total clearance of the analyte in serum following IV infusion (CL)
Vss | from 0 to day 99
  • Volume of distribution at steady state (Vss)
Vz | from 0 to day 99
  • Volume of distribution during the terminal phase λz following an intravascular dose (Vz)
Immunogenicity | from 0 to day 99
  Incidence of anti drug antibodies (ADAs), including neutralizing ADAs (NADAs)

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, M.D., Principal Investigator — The First Hospital of Jilin University; Chen Yu, M.D., Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Zhu X, Qian H, Sun J, Wu M, Yu C, Ding Y, Zhang X, Chai K, Li X. A phase 1 randomized study compare the pharmacokinetics, safety and immunogenicity of HLX04 to reference bevacizumab sourced from the United States, the European Union, and China in healthy Chinese male volunteers. Cancer Chemother Pharmacol. 2021 Sep;88(3):465-474. doi: 10.1007/s00280-021-04297-z. Epub 2021 Jun 4. PMID 34086067
- See also: Related Info — https://doi.org/10.1093/annonc/mdy431.019